CLINICAL TRIAL: NCT03276182
Title: Evaluation of Meibomian Gland Dysfunction Before and After Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2015-0851
Record Dates: First submitted 2017-08-29; First posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-08

CONDITIONS: Cataract Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cataract patients (Experimental): cataract patients undergoing phacoemulsification
  Interventions: Device: Lipiview 2

INTERVENTIONS:
Device: Lipiview 2 — Tear film lipid layer thickness and meibomian gland dropout were measured by LipiView interferometer (TearScience Inc, Morrisville, NC)

SUMMARY:
This study will compare cataract patients before and after phacoemulsification. Evaluations will be performed before and 1 and 3 months following cataract surgery, including parameters of dry eye syndrome and MGD. Dry eye syndrome parameters included TBUT, Schirmer's test type I, Oxford staining score, and the Ocular Surface Disease Index (OSDI) Questionnaire. MGD parameters consisted of lipid layer thickness (LLT), lid margin abnormality, meibum quality, meibum expressibility, MG orifice obstruction, MGD stage, and MG dropout.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cataract surgery planning with phacoemulsification and intraocular lens implantation with or without mild dry eye syndrome

Exclusion Criteria:

* the previous use of eye drops, except artificial tears within 3 months before cataract surgery
* a history of previous ocular surgery or trauma
* the presence of ocular comorbidities such as glaucoma, uveitis, cystoid macular edema, and any surgical complications including rupture of the posterior capsule during cataract surgery.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
the change of parameters associated with dry eye syndrome | baseline and 1 month after POD(postoperative day)
  Analysis the change of parameters associated with dry eye syndrome before and after cataract surgery measured by lipiview 2.
the change of parameters associated with meibomiangland dysfunction | baseline and 1 month after POD(postoperative day)
  Analysis the change of parameters associated with meibomiangland dysfunction before and after cataract surgery measured by lipiview 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No